CLINICAL TRIAL: NCT02928419
Title: Efficacy of Eltrombopag Plus Lenalidomide Combination Therapy in Patients With IPSS Low and Intermediate-risk Myelodysplastic Syndrome With Isolated del5q: a Multicenter, Randomized, Double-blind, Placebo Controlled Study - QOL-ONE Rev2MDS
Brief Title: Efficacy of Eltrombopag Plus Lenalidomide Combination Therapy in Patients With IPSS Low and Intermediate-risk Myelodysplastic Syndrome With Isolated del5q
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: "the study has been closed due to a low rate of patient enrollment (2 patients since the start of the trial)"
Sponsor: Associazione Qol-one (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QOL-ONE Rev2MDS
Record Dates: First submitted 2016-10-05; First posted 2016-10-10 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — eltrombopag; Lenalidomide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Eltrombopag) (Experimental): Arm 1 is the active treatment arm
  Interventions: Drug: Eltrombopag/Revolade; Drug: Lenalidomide
- Arm 2 (Placebo) (Placebo Comparator): Arm 2 is the control arm
  Interventions: Other: Placebo; Drug: Lenalidomide

INTERVENTIONS:
Drug: Eltrombopag/Revolade — From day 1, patients presenting with PLT counts ≤ 100 Gi/L at any time will receive oral eltrombopag for a maximum of 36 months.
  Starting dose will depend on PLT count determined on the day of first dose of eltrombopag. For patients experiencing PLT count 70 to 100 Gi/L, initial dosing is 50 mg/day. For subjects presenting with PLT counts < 70 Gi/L initial dosing is 100 mg/day. The dose of study medication must be increased sequentially by 50 mg every 7 days, up to a maximum dose of 300 mg/day until PLT ≥ 100 Gi/L. For East Asian subjects, a maximum dose of 150 mg is permitted.
  Arms: Arm 1 (Eltrombopag)
Other: Placebo — From day 1, patients presenting with PLT counts ≤ 100 Gi/L at any time will receive oral placebo for a maximum of 36 months.
  Starting dose will depend on PLT count determined on the day of first dose of placebo. For patients experiencing PLT count 70 to 100 Gi/L, initial dosing is 50 mg/day. For subjects presenting with PLT counts < 70 Gi/L initial dosing is 100 mg/day. The dose of study medication must be increased sequentially by 50 mg every 7 days, up to a maximum dose of 300 mg/day until PLT ≥ 100 Gi/L. For East Asian subjects, a maximum dose of 150 mg is permitted.
  Arms: Arm 2 (Placebo)
Drug: Lenalidomide — All patients will receive oral lenalidomide 10 mg/day for 21 days every 28 days. Patients will receive lenalidomide dosing according to the lenalidomide product information. Patients obtaining an erythroid response according to IWG 2006 criteria within the first 24 weeks will continue lenalidomide treatment until progression or other reasons for permanent discontinuation

SUMMARY:
Myelodysplastic syndromes (MDS) prevail in elderly patients and are characterized by inefficient erythropoiesis and peripheral cytopenias. Supportive care still represents the main therapeutic option in most patients. Quality of life is deteriorated mostly by anemia and by limitations due to dependence on transfusions, thrombocytopenia, and neutropenia. The only treatment available for severe thrombocytopenia consists of PLT transfusions, mainly in the presence of bleeding.

In patients with low and intermediate-1 risk MDS with an isolated deletion 5q cytogenetic abnormality, red blood cell (RBC) transfusion-dependence is a prevalent condition. For these latter patients reaching transfusion-dependence, lenalidomide, an immunomodulatory drug, has been approved by FDA and EMA. It has been shown that the drug induces significant erythroid (about 65%) and cytogenetic responses which have been associated with a survival benefit. In patients with MDS with del5q and serum erythropoietin levels > 500 miU/L, lenalidomide dosing of 10 mg/day for 21 days every 28, rather than 5 mg dosing, induces higher rates of transfusion-independence and cytogenetic responses with a trend to survival advantage. As a consequence, the recommended starting dose of lenalidomide is 10 mg orally once daily on days 1-21 of repeated 28-day cycles. Lenalidomide treatment must not be started if the Absolute Neutrophil Counts (ANC) < 0.5 Gi/L and/or PLT counts < 25 Gi/L.

For patients who are dosed initially at 10 mg and who experience thrombocytopenia < 25 Gi/L (45-75%), it is recommended to interrupt lenalidomide treatment until PLT count returns to ≥ 25 Gi/L on at least 2 occasions for ≥ 7 days or when the PLT count recovers to ≥ 50 Gi/L at any time, to resume lenalidomide at 50% dose reduction.

Eltrombopag is an orally bioavailable agonist of the thrombopoietin receptor. It has been shown that in patients affected by MDS and by acute myeloid leukemia, Eltrombopag neither increases the proliferation, nor the clonogenic growth capacity of bone marrow blasts. Furthermore, Eltrombopag induces an increase in the megakaryocytic differentiation and in the formation of normal megakaryocytic colonies. These results provide the rationale for pursuing further research on Eltrombopag for the treatment of thrombocytopenia in case of MDS.

Preliminary results of an ongoing randomized trial, EQoL-MDS, for the evaluation of efficacy, safety of eltrombopag for thrombocytopenia of low and intermediate-1 IPSS risk MDS has shown that eltrombopag is able to significantly raise PLT counts in about 65% of patients without additional toxicity Furthermore, the combination of lenalidomide and eltrombopag resulted in significant inhibitory effects on the growth of leukemic colonies in the majority of primary MDS and AML samples. Most importantly, eltrombopag was able to reverse the anti-megakaryopoietic effects of lenalidomide in primary MDS patient samples. These results provide a preclinical rationale for the use of this combination in MDS and AML

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (18 years of age or older) with MDS and low or intermediate-1 IPSS risk and del5q as a single abnormality, at the time of their screening and enrollment into the study
* Subjects must not have received any prior treatment course with any immunomodulating agent nor TPO-R agonists
* Subjects must be dependent on regular packed RBC transfusions, as defined by international working group 2006 criteria, and must have a PLT count taken within the 4 weeks prior to screening that is >25 Gi/L.
* Absolute Neutrophil Counts (ANC) ≥ 0.5 GiL
* Resistant or refractory to erythropoetic stimulating agents (ESAs) and/or serum erythropoetin levels > 500 miU/L
* Subjects must be ineligible or relapsed or refractory to receive treatment options of azacitidine and decitabine.
* Subjects must have PLT count and RBC and PLT transfusion data available over a period of 8 weeks prior to screening.
* During the 2 months prior to randomization, subjects must have a baseline BM examination including all of the following: cytomorphology, cytogenetics and histology
* ECOG Performance Status must be 0-3.
* The following clinical chemistries MUST NOT exceed the upper limit of normal (ULN) reference range: creatinine, ALT, AST, total bilirubin (except for Gilbert's Syndrome), gamma-gt and alkaline phosphatase. In addition, albumin must not be below the lower limit of normal (LLN) by more than 10%.
* If subject meets the criteria for childbearing potential:

  1. Negative pregnancy test in female subjects within the 3 days prior to Day 1 of 1st cycle and effective contraception for at least 4 weeks.
  2. Subject is practicing an acceptable method of contraception (documented in chart). Female subjects (or female partners of male subjects) must either be of non-childbearing potential (hysterectomy, bilateral oophorectomy, bilateral tubal ligation or post-menopausal >1 year), or of childbearing potential and use of an highly effective method of contraception from 2 weeks prior to administration of study medication, throughout the study, and 28 days after completion or premature discontinuation from the study.
* Criteria for women of non-childbearing potential: A female patient or a female partner of a male patient is considered to have childbearing potential unless she meets at least one of the following criteria:

  1. Age ≥ 50 years and naturally amenorrhoeic for ≥ 1 year (amenorrhoea following cancer therapy or during lactation does not rule out childbearing potential).
  2. Premature ovarian failure confirmed by a gynaecologist
  3. Previous bilateral salpingo-oophorectomy, or hysterectomy
  4. XY genotype, Turner syndrome, uterine agenesis.
* Subject is able to understand and comply with protocol requirements and instructions.
* Subject has signed and dated informed consent.

Exclusion Criteria:

* MDS with intermediate-2 or high IPSS risk
* Additional cytogenetic abnormalities
* Transfusion independence (TI) by IWG 2006 criteria
* Absolute Neutrophil Count < 0.5 Gi/L and/or Platelet counts < 25 Gi/L
* History of treatment for cancer with systemic chemotherapy and/or radiotherapy within the last 2 years
* History of treatment with immunomodulatory drugs or other TPO-R agonists.
* Thrombophilia, pre-existing history of thrombosis, cardiovascular disease (including congestive heart failure, New York Heart Association [NYHA] Grade III/IV), or arrhythmia known to increase the risk of thromboembolic events (e.g. atrial fibrillation), or subjects with a QTc >450 msec (QTc >480 msec for subjects with Bundle Branch Block)
* Bone Marrow fibrosis that leads to an inability to aspirate marrow for assessment.
* Leukocytosis >=25,000/uL prior to Day 1 of study medication.
* Monocytosis > 1000/ uL prior to Day 1 of study medication.
* Female subjects who are nursing or pregnant (positive serum or urine Beta-human chorionic gonadotropin [B-hCG] pregnancy test).
* Women of childbearing potential unless all of the conditions of the Pregnancy Prevention Programme illustrated in sections 6.4 are met (see sections 6.4).
* Known hypersensitivity to lenalidomide.
* Current alcohol or drug abuse.
* Treatment with an Investigational Product within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication.
* Active and uncontrolled infections.
* Subjects infected with Hepatitis B, C or Human Immunodeficiency Virus (HIV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-05; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Response (patients number with composite endpoint experience) | 24 weeks
  To evaluate the effect of eltrombopag treatment relative to placebo on the incidence of the "composite endpoint" (PLT<25 Gi/L or bleeding event with WHO bleeding score >1 or study discontinuation), in the first 24 weeks, after experiencing PLT<100 Gi/L

SECONDARY OUTCOMES:
Response (patients number with composite endpoint experience on long-term) | 36 months
  The composite endpoint during the entire study period
Safety (number of adverse events) | 36 months
  Safety and tolerability in terms of frequency of adverse events (AE)s and serious adverse events (SAE).
Cytogenetic responses | 36 months
  Proportion of cytogenetic responses, according to IWG 2006 criteria
Duration of cytogenetic response | 36 months
  Duration of cytogenetic response
Hb changes | 24 weeks
  Hb changes within the first 24 weeks.
Erythroid response | 36 months
  Erythroid response, transfusion-independence (TI) and duration of TI.
Quality of Life (QOL) | 36 months
  Changes in QOL scores
Progression free survival | 36 months
  Progression free survival from baseline
Overall survival | 36 months
  Overall survival from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Esther Natalie Oliva, MD, Study Chair — QOL-ONE Associazione Culturale e di Ricerca
Locations (50):
- France (14):
  - CHU d'Angers, Angers
  - Centre Henri Mondor, Créteil
  - CHU de Grenoble, Grenoble
  - Centre Le Mans, Le Mans
  - CHRU de Limoges, Limoges
  - Centre Hospitalier Lyon Sud, Lyon
  - Centre de Marseille, Marseille
  - CHU Brabois, Nancy
  - Centre de Nantes, Nantes
  - Hopital Archet 1, Nice
  - Centre Hospitalier Universitaire de Nimes, Nîmes
  - Centre de Rouen, Centre Henri Becquerel, Rouen
  - CHU Purpan, Toulouse
  - CHU de Bretonneau, Tours
- Greece (7):
  - "G.Gennimatas" General Hospital of Athens, Athens
  - University Hospital "Atticon",, Athens
  - University Hospital "Laikon", Athens
  - University Hospital of Crete, Crete
  - University Hospital of Larissa, Larissa
  - University Hospital of Patras, Pátrai
  - "George Papanicolaou General Hospital of Thessaloniki, Thessaloniki
- Italy (29):
  - A.O. SS. Antonio e Biagio e Cesare Arrigo, Alessandria, AL
  - Ospedale Riuniti, Ancona, AN
  - Ospedale Cardinal Massaia, Asti, AT
  - A.O. S. Giovanni Moscati, Avellino, AV
  - Presidio Ospedaliero Oncologico Businco, Cagliari, CA
  - Ospedale L'Annunziata, Cosenza, CS
  - Ospedale Ferrarotto, Catania, CT
  - Ospedale Garibaldi, Catania, CT
  - Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, FG
  - Azienda Ospedaliera Universitaria Careggi, Florence, FI
  - Ospedale Vito Fazzi, Lecce, LE
  - A.O. San Gerardo, Monza, MB
  - IRCCS Ospedale Maggiore Policlinico, Milan, MI
  - Ospedale Niguarda, Milan, MI
  - Ospedale Civile Spirito Santo, Pescara, PE
  - Azienda Ospedaliera Bianchi-Melacrino-Morelli, Reggio Calabria, RC
  - Arcispedale di Santa Maria Nuova, Reggio Emilia, RE
  - A.O. San Camillo Forlanini, Roma, RM
  - Ospedale Sant'Eugenio, Roma, RM
  - Policlinico Agostino Gemelli, Roma, RM
  - Azienda Ospedaliera Sant'Andrea, Rome, RM
  - IRCCS Istituto Regina Elena, Rome, RM
  - Ospedale Nuova Regina Margherita, Rome, RM
  - Policlinico Umberto I, Rome, RM
  - Policlinico Universitario Tor Vergata, Rome, RM
  - Policlinico Santa Maria alle Scotte, Siena, SI
  - A.O. Santa Maria, Terni, TE
  - A.O. Citta' della Salute e della Scienza di Torino, Torino, TO
  - U.O. Citta' della Salute e della Scienza di Torino, Torino, TO

IPD SHARING:
Plan to Share IPD: Undecided